CLINICAL TRIAL: NCT06098352
Title: The Impact of a Continuous Performance Task on the Stress Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Redlands (Other)
Responsible Party: Principal Investigator, Lisa Olson, Professor of Biology, University of Redlands
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2013-31-REDLANDS
Record Dates: First submitted 2023-10-18; First posted 2023-10-24 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Stress
Keywords: stress; anxiety; blood pressure; skin conductance level; heart rate variability; attention
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: All participants will be measured at baseline and then during an attention task.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PEBL Continuous Performance Task (Experimental): Participants will take the PEBL Continuous Performance Task, a 14 minute attention test requiring participants to press the space bar when certain letters are shown on the screen.
  Interventions: Behavioral: PEBL Continuous Performance Task

INTERVENTIONS:
Behavioral: PEBL Continuous Performance Task — A PEBL version of the Conners Continuous Performance Task
  Other Names: Conners Continuous Performance Task

SUMMARY:
The goal of this clinical trial is to learn about the impact of taking a continuous performance attention test on the physiological stress response in college students. The main questions it aims to answer are:

* Does taking an attention test cause participants to have increases in heart rate, blood pressure, and sweat?
* Does taking an attention test cause participants to have a decrease in heart rate variability?
* Are there relationships between participants' levels of anxiety, perceived stress, and mindfulness to their physiological changes?

Participants will

* Answer questionnaires about anxiety, stress, and mindfulness
* Have baseline measurements taken for blood pressure, sweat, and heart rate variability
* Take the PEBL Continuous Performance Task (a 14 minute attention test) while having the measurements listed above taken again

DETAILED DESCRIPTION:
The PEBL Continuous Performance Task is an example of a mental stressor which requires vigilance and effort. We hypothesize that a sympathetic nervous system response will be evident in comparing physiological parameters during the attention task versus the preceding resting baseline period. Exploratory analyses will assess relationships between psychological measures of anxiety, stress, and mindfulness with this physiological response and the number of errors on the attention test.

ELIGIBILITY:
Inclusion Criteria:

* English language proficiency
* First year, first semester student enrolled in Students Together Empowering Peers course at the University of Redlands

Exclusion Criteria:

* severe mental health issues
* currently taking anti-anxiety medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-09-17 (Actual); Primary Completion 2013-09-25 (Actual); Study Completion 2013-09-25 (Actual)

PRIMARY OUTCOMES:
Blood pressure | Measured once after an 8 minute resting baseline, then 2 minutes into the attention task, and 10 minutes into the attention task. Data collection was then complete.
  Systolic and diastolic
Skin conductance level | Measured continuously during an 8 minute resting baseline, then continuously for the 14 minute attention task. Data collection was then complete.
  levels of sweat due to sympathetic nervous system activation
Heart rate variability | Measured continuously during an 8 minute resting baseline, then continuously for the 14 minute attention task. Data collection was then complete.
  Normalized high frequency HRV

SECONDARY OUTCOMES:
State Trait Anxiety Inventory (STAI) | Questionnaire completed on day of enrollment (<30 minutes)
  Spielberger, C.D., R.L. Gorsuch, and R.E. Lushene, 1970. Scores on each of the state and trait sections range from 20 (low anxiety) to 80 (high anxiety)
Perceived Stress Scale (PSS-10) | Questionnaire completed on day of enrollment (<30 minutes)
  Cohen, S., T. Kamarck, and R. Mermelstein. Journal of Health and Social Behavior, 1983. Scores range from 0 (low perceived stress) to 40 (high perceived stress)
Mindful Awareness and Attention Scale (MAAS) | Questionnaire completed on day of enrollment (<30 minutes)
  Brown, K.W. and R.M. Ryan. Journal of Personality and Social Psychology, 2003. Scores range from 1 (least mindful) to 6 (most mindful)
PEBL Continuous Performance Task Foil Accuracy Rate | 14 minute attention task on the day of the experiment
  For trials where participants were presented with a foil, the percent in which the participant did not commit a commission error (participant correctly did not press spacebar). Ranges from 0 - 100% accuracy.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa E Olson, Ph.D., Principal Investigator — University of Redlands
Locations (1):
- University of Redlands, Redlands, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized participant data will be provided upon request
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Starting after publication, and up to 10 years after publication
Access Criteria: Will be provided to researchers affiliated with an academic institution upon request

REFERENCES:
- [Background] Brown KW, Ryan RM. The benefits of being present: mindfulness and its role in psychological well-being. J Pers Soc Psychol. 2003 Apr;84(4):822-48. doi: 10.1037/0022-3514.84.4.822. PMID 12703651
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Spielberger, C.D., R.L. Gorsuch, and R.E. Lushene, Manual for the state-trait anxiety inventory. 1970: Consulting Psychologists Press, Palo Alto, CA.
- [Background] The PEBL Project. (2019). PEBL. Retrieved from https://pebl.sourceforge.net
- [Derived] Bautista BR, Gurning J, Marks M, Ortyn D, Salinas R, Olson LE. The sympathetic nervous system response to a Continuous Performance Task. MicroPubl Biol. 2024 Jun 12;2024:10.17912/micropub.biology.001059. doi: 10.17912/micropub.biology.001059. eCollection 2024. PMID 38938412